CLINICAL TRIAL: NCT04671134
Title: Evaluation of State and Shade of White Spot Lesions After Using Different Remineralizing Agents (An in Vivo Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hany Helmy Elsayed Mohammed, Principle Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 581/3287
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: White Spot Lesion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biomimetic remineralizing agent (Experimental)
  Interventions: Other: Biomimetic remineralizing agent; Other: Resin Modified Glass Ionomer Varnish
- Resin modified glass ionomer varnish (Active Comparator)
  Interventions: Other: Biomimetic remineralizing agent; Other: Resin Modified Glass Ionomer Varnish

INTERVENTIONS:
Other: Biomimetic remineralizing agent — Self-assempling peptide
Other: Resin Modified Glass Ionomer Varnish — Resin Modified Glass Ionomer Varnish

SUMMARY:
The aim of the study is to evaluate the effect of Biomimetic remineralizing agent and resin modified glass ionomer varnish on color shade and state of white spot lesions immediately, after 3 months, and after 6 months. (An in vivo study).

ELIGIBILITY:
Inclusion Criteria:

1. Patients included in this clinical trial were less than 30 years old.
2. Patients with good general health.
3. Patients who will agree to the consent and will commit to follow-up period.
4. Fully erupted anterior teeth with no cavitated lesions.

Exclusion Criteria:

1. Patients with any systemic disease that may affect normal healing.
2. Patient with bad oral hygiene.
3. Tetracycline or florosis staining.
4. Patients who could/would not participate in all times of follow-up.
5. Untreated periodontal disease was not allowed.
6. Active caries or defective Restorations in 6 anterior teeth.
7. Bleaching history
8. Patients participating in more than 1 dental study.
9. Patient received fluoride varnish before.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
state of lesions | 6 months.
  Digital scores

SECONDARY OUTCOMES:
shade of lesions | 6 months
  Digital scores

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR